CLINICAL TRIAL: NCT01165515
Title: Endostatin Serum Levels During Bicycle Stress Test in Different Samples
Brief Title: Endostatin Serum Levels During Bicycle Stress Test
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Jeanette Strametz-Juranek, Ao.Univ.Prof.Dr, Medical University of Vienna
Other Study IDs: 220/2007
Record Dates: First submitted 2010-07-13; First posted 2010-07-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Smoking; Cardiac Diseases
MeSH Terms: conditions — Smoking; Heart Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (13):
- Healthy young females: 20 healthy females, aged between 18 and 35 years
- Healthy young males: 20 healthy males, aged between 18 and 35 years
- Healthy elderly smokers: 20 healthy smokers, aged between 45 and 75 years
- Healthy elderly non-smokers: 20 healthy non-smokers, aged between 45 and 75 years
- Healthy young female smokers: 20 healthy female smokers, aged between 18 and 35 years
- Healthy young male smokers: 20 healthy male smokers, aged between 18 and 35 years
- Healthy postmenopausal women: 20 healthy postmenopausal women
- Female CMP Patients: 20 female patients suffering from cardiomyopathy (ischemic or dilating)
- Male CMP Patients: 20 male patients suffering from cardiomyopathy (ischemic or dilating)
- Female CHD patients: 30 female patients suffering from cardiac heart disease, before aorto-coronary bypass surgery (and after)
- Male CHD Patients: 30 male patients suffering from cardiac heart disease, before aorto-coronary bypass surgery (and after)
- male athlets: 20 male athlets
- female athlets: 20 female athlets

SUMMARY:
Endostatin, a 20-kDa cleavage product of collagen XVIII, is a component of the extracellular matrix expressed in the basement membrane. As a potent inhibitor of angiogenesis, endostatin induces endothelial cell apoptosis and diminishes cell migration, adhesion and proliferation.

Endostatin may stop the progression of atherosclerosis. Atherosclerotic heart disease involves unwanted tissue growth. By cutting off the blood supply from a plaque the likelihood of plaque rupture may eventually be reduced. Recent data indicates that the loss of collagen XVIII/endostatin is related to the enhancement of neo-vascularization and vascular permeability in atherosclerosis. Plaque neo-vascularization strongly correlates with the regional content of inflammatory cells. Furthermore, increased vascular permeability enhances lipid accumulation in the vessel walls, hence increasing foam cells.

Therapeutic angiogenesis is a most promising strategy for the treatment of myocardial infarction. However, it remains unknown if and how endogenous angiogenesis inhibitors, such as endostatin, regulate angiogenesis in myocardial infarction. Rat models showed that after myocardial infarction endostatin neutralization displayed adverse left ventricular remodeling and severe heart failure compared with controls. Although angiogenesis was increased, tissue remodeling and interstitial fibrosis were further exaggerated in post-myocardial infarction hearts by endostatin neutralization.

However, several studies suggest that endostatin may locally modulate coronary collateral formation by inhibiting collateral vessel formation in patients with ischemic heart disease.

During treadmill exercise tests in healthy volunteers a significant increase in circulating endostatin levels can be observed. Exercise induces angiogenesis in cardiac and skeletal muscles by decreasing endostatin in the muscle tissues to increase blood flow to these metabolically active tissues. Thereby endostatin is released into the general circulation.

In summary, endostatin might be a new weapon to fight against atherosclerotic progression by inhibiting neo-vascularization of atherosclerotic plaques.

ELIGIBILITY:
Inclusion Criteria:

* Smoking/Non smoking
* Healthy/non healthy (if for CMP, CHD study)
* Age (depending on the group affiliation)

Exclusion Criteria:

* Suffering from grave diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 patients, divided into sub-groups, always both genders will be tested for different conditions (smoking, age, CMP, CHD,...)
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2008-01; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Endostatin | baseline/maximum
  baseline sample will be drawn at rest; a second sample will be drawn 5 minutes after each individual reaches its peak workload (average time 10 minutes)

SECONDARY OUTCOMES:
catecholamine | baseline
  baseline sample will be drawn at rest
hemodynamic parameters | baseline
  heart rate and blood pressure behavior will be monitored throughout the entire bicycle stress test
catecholamine | day 1
  a second sample will be drawn 5 minutes after each individual reaches its peak workload (average time 10 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Strametz-Juranek, MD, Principal Investigator — MUV, Department of Internal Medicine II, Division of Cardiology
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Result] Sponder M, Dangl D, Kampf S, Fritzer-Szekeres M, Strametz-Juranek J. Exercise increases serum endostatin levels in female and male patients with diabetes and controls. Cardiovasc Diabetol. 2014 Jan 6;13:6. doi: 10.1186/1475-2840-13-6. PMID 24393402